CLINICAL TRIAL: NCT01295073
Title: Trientine Hydrochloride for the Prevention of Macular Edema After Cataract Surgery in Patients With Type 2 Diabetes Mellitus
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: appropriate study medication supply could not be identified
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, David Maberley, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H11-00165
Record Dates: First submitted 2011-02-10; First posted 2011-02-14 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Macular Edema Following Cataract Surgery
Keywords: Trientine; Cataract surgery; Macular Edema
MeSH Terms: conditions — Macular Edema | interventions — Trientine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Oral Trientine 1500mg x 1 week before cataract surgery and 3 days post surgery
  Interventions: Drug: Trientine Hydrochloride
- B (Placebo Comparator): Oral Placebo x 1 week before cataract surgery and 3 days post surgery
  Interventions: Other: For Arm B there is no therapeutic intervention other than standard of care, which is cataract surgery.

INTERVENTIONS:
Drug: Trientine Hydrochloride — Arm A's therapeutic intervention is the use of Trientine Hydrochloride for 10 days in the perioperative period.
  All participating subjects will all receive cataract surgery according to present standards of care; however, subjects randomized the intervention group (trientine hydrochloride) will be on a 10 day course of oral Trientine at 1500mg administered for 7 days prior to and 3 days after surgery.
  Other Names: Syprine
  Arms: A
Other: For Arm B there is no therapeutic intervention other than standard of care, which is cataract surgery. — see above
  Arms: B

SUMMARY:
The primary purpose of the protocol is to evaluate whether Trientine Hydrochloride, a copper chelator which is an agent that binds with and removes copper, will be effective in minimizing macular edema after cataract surgery in individuals with type 2 diabetes. It is our hypothesis that there will be a reduction in copper-attributed inflammation after surgery resulting a decrease in edema.

DETAILED DESCRIPTION:
Individuals with type II Diabetes Mellitus who present to the UBC/VGH Eye Care Centre for cataract surgery will be offered participation in this study. Cataract surgery will be performed according to the surgeons' normal protocols and the present standards of care; however, subjects will be randomized to either a 10-day course of oral Trientine at 1500mg/day administered for 7 days prior to and 3 days after the surgery, or to placebo. Urinary copper levels will be evaluated before and after Trientine administration to determine the efficacy of copper chelation at the time of surgery.

Baseline ocular exams, bloodwork and urine collection will be organized or performed at the two screening visits up to two months before the date of cataract surgery according to the research protocol (flowsheet included at the end). Subjects will also be evaluated at Day1 post-operative, Day 7 (Week #1) post operative, and Day 28-30 (Month 1)post operative with Ocular Coherence Tomography (retinal thickness measurements). Fundus photography and visual acuity testing will be done at Screening and month 1. A final phlebotomy to rule out copper deficiency anemia will be required at month 1 as well.

ELIGIBILITY:
INCLUSION CRITERIA:

1. A diagnosis of type 2 Diabetes Mellitus.
2. Early Treatment of Diabetic Retinopathy Study (ETDRS) eye chart score of 34 to 73 letters at 2 meters following auto-refraction. (20/20 to 20/320 [logMAR 0 to 1.2] for study eye.
3. Willing and able to participate and provide written informed consent.
4. Must be 19 years of age or older
5. Patients must require cataract surgery as determined by an ophthalmologist.
6. Patients must have standard, uncomplicated cataract surgery with a foldable lens planned.

EXCLUSION CRITERIA:

1. Individuals with active retinal neovascularization.
2. Any intraocular surgery within 2 months or laser surgery within 1 month in the study eye.
3. Prior retinal or vitreous surgery including posterior segment vitrectomy or scleral buckling.
4. Inadequate initial OCT scan for reliable baseline measurement of retinal thickness.
5. Current macular edema not related to diabetes.
6. Patients who have received treatment with Avastin or Lucentis or laser in either eye in the last 3 months.
7. Other ocular disease unrelated to diabetes or cataract that the investigator believes could be affect macular imaging or visual outcome.
8. Medical conditions requiring constant use of mineral supplements (copper, iron or zinc in particular). This does not include those with Age-related Macular Degeneration (AMD) who may safely stop vitamins and minerals for the 10 day course of the treatment.
9. Patients with anemia.
10. Patients with physical or mental disabilities that prevent accurate testing.
11. Active hepatitis, clinically significant liver disease, or a recent history of alcohol abuse.
12. Any evidence of renal failure or an eGFR of less than 80% of age-adjusted normals.
13. Patients who had a stroke or myocardial infarction within the preceding 6 months or who have ventricular tachycardia under treatment.
14. History of severe cardiac disease or unstable angina.
15. Subjects who are in an experimental therapy study or who have received experimental therapy within the last 12 weeks.
16. Subjects who are a poor medical risk because of other systemic diseases or active uncontrolled infections.
17. Subjects with inflammatory systemic diseases, such as systemic lupus erythematous.
18. Women of childbearing potential not on 2 effective forms of birth control.
19. Women who are pregnant or plan to become pregnant.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Change in retinal thickness measurements by Optical Coherence Tomography (OCT) from screening to Day 28 between subjects undergoing surgery with and without Trientine use. | Screening, Day 28

SECONDARY OUTCOMES:
Secondary analyses will involve evaluations of the change in visual acuity and fundus photography results from screening to Day 28. | Screening, Day 28

CONTACTS AND LOCATIONS:
Overall Officials: David Maberley, MD,FRCSC,MSc(Epid), Principal Investigator — University of British Columbia
Locations (1):
- Univeristy of British Columbia/Vancouver Coastal Health Authority - Eye Care Center, Vancouver, British Columbia, Canada